CLINICAL TRIAL: NCT00005333
Title: Epidemic Hypertension in Nigerian Workers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4188; R01HL044413 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
Originally from 1991 to 1991, to test the hypothesis that differences in hypertension prevalence in Nigerian workers were primarily related to differences in socioeconomic status (SES). At renewal in 1996, to determine the importance of weight gain and weight-related factors in blood pressure.

DETAILED DESCRIPTION:
BACKGROUND:

This dynamic population provided a valuable opportunity to gain important information about the etiology of hypertension which would be much more difficult to gain from a United States Black population because higher weight and blood pressure are already entrenched and static in the United States population.

DESIGN NARRATIVE:

From 1991 to 1996, a cross-sectional study was conducted to test the hypothesis that differences in hypertension prevalence were primarily related to differences in SES. The higher prevalence of hypertension among the high SES Nigerian professionals was thought to be related to higher weight, caloric intake, Westernization of diet, alcohol intake, sodium intake, cardiovascular reactivity, and stress due to job, migration, and change in SES, and to reduced potassium intake and physical activity. Civil servants were systematically sampled from civil service employee lists. Data were collected on blood pressure; urinary sodium, potassium, and protein; diet; anthropometry; electrocardiogram; serum insulin; stress in the work environment, migration history, and cardiovascular reactivity.

In FY 1992, the Office of Research on Women's Health provided supplemental funds to enlarge the study and to perform gender analyses. The supplemental funds were used to determine whether fatty acid distributions, and their relationships to cardiovascular risk factors differed between Nigerian women and United States Black women; United States Black women and United States white women; and Nigerian women and Nigerian men. Forty men and forty women, ages 18 to 30, were chosen randomly from the Nigerian civil servant population. Subjects with hypertension, those using oral contraceptives, or any medication affecting the sympathetic nervous system, were excluded. The Nigerian subjects were compared with 40 Black and 40 white healthy female volunteers at the University of Pittsburgh.

The grant was renewed in 1996 through August 2001 to conduct a longitudinal study of 726 members of the original cohort. The purpose was to determine the importance of weight gain and weight-related factors, and the possible interaction of other factors, e.g. psychosocial, electrolytes, reactivity, macronutrient intake, to change in blood pressure. Factors related to weight gain were identified. The high prevalence of the electrocardiogram left ventricular hypertrophy (ECG-LVH) was validated against echocardiographic measures (ECHO-LVH). Predictors of change in ECG-LVH, and the correlates of microalbuminuria were identified. In Year 2 (Cohort Year 4) half of the population was restudied with echocardiography, cardiovascular reactivity, and new psychosocial measures. In Year 4 (Cohort Year 6), with the exception of cardiovascular reactivity, the full cohort was re-examined for baseline measures, including multiple blood pressure readings, height, weight, waist, hips, ECG, physical activity, two 24 hour dietary recalls, alcohol intake, menopausal status, psychosocial measures, 24 hour urine for sodium, potassium, creatinine, micro-albuminuria, and fasting serum for lipids, insulin, glucose, and creatinine.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-01; Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clareann Bunker — University of Pittsburgh

REFERENCES:
- [Background] Evans RW, Bunker CH, Ukoli FA, Kuller LH. Lipoprotein (a) distribution in a Nigerian population. Ethn Health. 1997 Mar-Jun;2(1-2):47-58. doi: 10.1080/13557858.1997.9961814. PMID 9395588
- [Background] Yeh LL, Kuller LH, Bunker CH, Ukoli FA, Huston SL, Terrell DF. The role of socioeconomic status and serum fatty acids in the relationship between intake of animal foods and cardiovascular risk factors. Ann Epidemiol. 1996 Jul;6(4):290-8. doi: 10.1016/s1047-2797(96)00023-3. PMID 8876839
- [Background] Bunker CH, Ukoli FA, Okoro FI, Olomu AB, Kriska AM, Huston SL, Markovic N, Kuller LH. Correlates of serum lipids in a lean black population. Atherosclerosis. 1996 Jun;123(1-2):215-25. doi: 10.1016/0021-9150(96)05810-8. PMID 8782852
- [Background] Markovic N, Matthews KA, Huston SL, Egbagbe E, Ukoli FA, Bunker CH. Blood pressure reactivity to stress varies by hypertensive status and sex in Nigerians. Am J Epidemiol. 1995 Nov 15;142(10):1020-8. doi: 10.1093/oxfordjournals.aje.a117554. PMID 7485046
- [Background] Bunker CH, Ukoli FA, Matthews KA, Kriska AM, Huston SL, Kuller LH. Weight threshold and blood pressure in a lean black population. Hypertension. 1995 Oct;26(4):616-23. doi: 10.1161/01.hyp.26.4.616. PMID 7558221
- [Background] Ukoli FA, Bunker CH, Fabio A, Olomu AB, Egbagbe EE, Kuller LH. Body fat distribution and other anthropometric blood pressure correlates in a Nigerian urban elderly population. Cent Afr J Med. 1995 May;41(5):154-61. PMID 7628000
- [Background] Markovic N, Olomu IN, Bunker CH, Huston SL, Ukoli FA, Kuller LH. Adequacy of a single visit for classification of hypertensive status in a Nigerian civil servant population. Int J Epidemiol. 1994 Aug;23(4):723-9. doi: 10.1093/ije/23.4.723. PMID 8002185
- [Background] Huston SL, Bunker CH, Ukoli FA, Rautaharju PM, Kuller LH. Electrocardiographic left ventricular hypertrophy by five criteria among civil servants in Benin City, Nigeria: prevalence and correlates. Int J Cardiol. 1999 Jul 1;70(1):1-14. doi: 10.1016/s0167-5273(99)00061-3. PMID 10402040
- [Background] Markovic N, Bunker CH, Ukoli FA, Kuller LH. John Henryism and blood pressure among Nigerian civil servants. J Epidemiol Community Health. 1998 Mar;52(3):186-90. doi: 10.1136/jech.52.3.186. PMID 9616424
- [Background] Desai PP, Bunker CH, Ukoli FA, Kamboh MI. Genetic variation in the apolipoprotein D gene among African blacks and its significance in lipid metabolism. Atherosclerosis. 2002 Aug;163(2):329-38. doi: 10.1016/s0021-9150(02)00012-6. PMID 12052480
- [Background] Forrest KY, Bunker CH, Kriska AM, Ukoli FA, Huston SL, Markovic N. Physical activity and cardiovascular risk factors in a developing population. Med Sci Sports Exerc. 2001 Sep;33(9):1598-604. doi: 10.1097/00005768-200109000-00025. PMID 11528351